CLINICAL TRIAL: NCT00909870
Title: A Prospective, Multi-Center, Randomized, Controlled Clinical Investigation of Dermagraft(R) in Subjects With Venous Leg Ulcers DEVO-Trial
Brief Title: Pivotal Trial of Dermagraft(R) to Treat Venous Leg Ulcers
Acronym: DEVO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABH-Dermagraft-001-08
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Venous Leg Ulcer
Keywords: Venous leg ulcer; randomized trial; clinical trial; Dermagraft; compression therapy; surgical debridement; venous stasis; chronic ulcer; chronic wound; fibroblasts
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Weekly applications of Dermagraft and compression dressings, in combination with systematic surgical wound debridement.
  Interventions: Device: Dermagraft(R)
- 2 (Active Comparator): Weekly application of compression dressings only, in combination with systematic surgical wound debridement.
  Interventions: Device: Profore

INTERVENTIONS:
Device: Dermagraft(R) — Weekly application of Dermagraft(R) with Profore compression as a secondary layer, in combination with systematic surgical wound debridement.
  Arms: 1
Device: Profore — Weekly application of Profore compression dressings, in combination with systematic surgical wound debridement.
  Arms: 2

SUMMARY:
This study randomly assigns patients with venous leg ulcers to receive standard therapy (compression) alone or compression plus Dermagraft(R). Dermagraft is a device containing live human fibroblasts grown on an absorbable Vicryl mesh. Patients are seen weekly until they heal or the 16-week treatment period is complete. Follow-up visits are conducted monthly for three months in order to assess patients for longer term safety.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* ABI > 0.80
* Three or fewer venous leg ulcers, if multiple must be separated by 2 cm
* Ultrasound demonstrates venous reflux >0.5 seconds
* Study wound present for 1-24 months
* Study wound 2-15 sq cm surface area
* Clean, granulating wound
* Patient able and willing to sign informed consent and comply with study procedures.
* Women of childbearing potential must use birth control pills, barriers or abstinence and have a negative pregnancy test.

Exclusion Criteria:

* Wound etiology uncertain or not from venous hypertension.
* BMI>40
* Acute or chronic infectious skin disease
* Allergy or intolerance to Profore(R)
* Wound infection, cellulitis, osteomyelitis
* >2 weeks' treatment with immunosuppressive agents in recent past
* Investigational drug use within 30 days
* Severe malnutrition, drug and/or alcohol abuse
* Malignant disease unless in remission for 5 years
* History of radiation at the study site
* Other conditions that could impede wound healing
* Known history of HIV or AIDS
* Prior participation in any Dermagraft study
* Treatment with other bioengineered tissue products within 30 days
* Unable to understand the aims and objectives of the trial
* Inability to comply with study protocol
* NYHA Class III or IV CHF
* Uncontrolled diabetes mellitus
* Dorsal foot ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Marston, MD, Principal Investigator — University of North Carolina School of Medicine, Chapel Hill, NC; Keith Harding, MD, Principal Investigator — Cardiff University School of Medicine, Wales, UK; David Bergqvist, MD, Principal Investigator — University of Uppsala, Sweden
Locations (70):
- United States (34):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Southern Arizona VA Health Care System (SAVAHCS), Tucson, Arizona
  - University of Arizona College of Medicine, Tucson, Arizona
  - Dr. Jagpreet S. Mukker, Fresno, California
  - VA Northern California Health Care System, Mather, California
  - Sutter Roseville Medical Center Wound Care Center, Roseville, California
  - Therapeutics Clinical Research, San Diego, California
  - General Vascular Surgery Group, San Leandro, California
  - Pacific Wound Center, Stockton, California
  - North American Center for Limb Preservation, New Haven, Connecticut
  - Providence Hospital, Washington D.C., District of Columbia
  - Foot & Ankle Associates of Florida, Altamonte Springs, Florida
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Comprehensive Wound Healing Center, Clearwater, Florida
  - Osceola Regional Wound Care Center, Kissimmee, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Doctor's Research Network, South Miami, Florida
  - Robert Snyder, DPM, CWS, Tamarac, Florida
  - Aiyan Diabetes Center, Evans, Georgia
  - Broadlawns Medical Center, Des Moines, Iowa
  - Boston Medical Center, Department of Vascular Surgery, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Covenant Wound Healing Center, Saginaw, Michigan
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - Overlook Hospital Wound Healing Program, Summit, New Jersey
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina Division of Vascular Surgery, Chapel Hill, North Carolina
  - Saint Vincent Health Center, Erie, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Jackson Madison County General Hospital, Jackson, Tennessee
  - Dixie Regional Meidcal Center, St. George, Utah
- Austria (2):
  - Private Practice FA fur Dermatologie Clinical Centre, Hartberg
  - Private Practice / Clinical Centre, Vienna
- East-Tallinn Central Hospital, Tallinn, Estonia
- Germany (2):
  - Dermatologische Gemeinschaftspraxis Professor Dr. med W. Vanscheidt, Freiburg im Breisgau
  - Germeinschaftspraxis Dres. Münter, Schiewe, Pohl Studienzentrum Dr. Münter, Hamburg
- Poland (12):
  - Institution DER-ART Scientific Research and Training Centre for Dermatosurgery, Gdynia
  - AKMed Medical Centre, Krakow
  - NZOZ Clinical for Vascular Diseases, Krakow
  - Malopolskie Centrum Medyczne, Krakow
  - 5 Wojskowy Szpital Kliniczny w Krakowie, Krakow
  - S. Zeromski Hospital Krakow, Krakow
  - NZOZ "Dermed" Medical Centre (Centrum Medyczne Sp. z.o.o.), Lodz
  - Clinical Trials Centre, Lublin
  - "NZOZ OPTI-MED Henryk Kaczmarek" Private Outpatient Clinic of Internal Medicine, Gastroenterology and Radiology, Nowy Sącz
  - "Medyk" Medical Center, Rzeszów
  - General Surgery Clinic Autonomous Public Central Clinical Hospital (SPCSK), Warsaw
  - NZOZ "Ars Medica" S.c. Wroclaw Health Centre (Wroclawskie Centrum Zdrowia), Wroclaw
- South Africa (13):
  - Langeberg Medical Centre, Kraaifontein, Cape Town
  - Worthwhile Clinical Trials Lakeview Hospital, Benoni, Johannesburg
  - Edenvale Hospital, c/o CEO Secretary, Edenvale, Johhanesburg
  - GCT-Mercantile Clinical Trial Centre, Korsten, Port Elizabeth
  - Synexus SA Watermeyer Clinical Research Centre, Meyerspark, Pretoria
  - Josha Research, Bloemfontein
  - Dr. D.R.Lakha, Private Practice, Johannesburg
  - I Engelbrecht Research, Lyttelton
  - Middelburg Hospital, Middelburg
  - Uncedo Clinical Research Services Mercantile Hospital, Port Elizabeth
  - Cachetmed Medical Centre, Potchefstroom
  - Randles Road Medical Centre, Sydenham, Durban
  - Clinical Projects Research SA, Worcester
- Sweden (2):
  - University of Lund Dept of Dermatology, Lund
  - Overlakare/Klinikchef Hud Kliniken, Stockholm
- United Kingdom (4):
  - Wound Clinic on Fairfield, Croydon, Surrey
  - Bradford Hospitals NHS Trust, Bradford
  - Cardiff University, Cardiff
  - Charing Cross Hospital, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening commenced in May 2009 and ended in November 2010.
  Study sites included vascular surgery, dermatology, and podiatry clinics.
  A total of 913 potential subjects were screened across 58 study centers; 395 subjects were screen failures.
  A total of 537 subjects were enrolled across 49 study centers.
Pre-assignment Details: Prior to study enrollment, all subjects signing informed consent proceeded through a two-week run-in phase in which all subjects received standard-of-care study ulcer treatment. During this phase, any subject not meeting inclusion/exclusion criteria was considered a screen failure and removed from the study.
Groups:
- Investigational Treatment (Dermagraft Plus Standard-of-Care): Weekly applications of Dermagraft and compression dressings, in combination with systematic surgical wound debridement.
- Active Control (Standard-of-Care): Weekly application of compression dressings only, in combination with systematic surgical wound debridement.
Period: Overall Study
Arm/Group | Investigational Treatment (Dermagraft Plus Standard-of-Care) | Active Control (Standard-of-Care)
Started | 274 | 263
Completed | 251 | 236
Not Completed | 23 | 27
Not completed — Adverse Event | 13 | 7
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 0 | 2
Not completed — Other | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Control (Standard-of-Care): Weekly application of compression dressings only, in combination with systematic surgical wound debridement.
- Total: Total of all reporting groups
Arm/Group | Investigational Treatment (Dermagraft Plus Standard-of-Care) | Control (Standard-of-Care) | Total
Number analyzed (Participants) | 274 | 263 | 537
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.1 (13.04) | 63.2 (14.46) | 63.1 (13.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 146 | 304
  Male | 116 | 117 | 233
Region of Enrollment [Number; unit: participants]
  United States | 94 | 93 | 187
  Estonia | 10 | 9 | 19
  Poland | 81 | 74 | 155
  South Africa | 73 | 71 | 144
  Germany | 8 | 8 | 16
  United Kingdom | 6 | 7 | 13
  Sweden | 2 | 1 | 3
Ulcer Size [Median (Full Range); unit: centimeters-squared] | 5.75 [1.5 to 19.3] | 5.90 [2.0 to 24.8] | 5.9 [1.5 to 24.8]
Ulcer Duration [Median (Full Range); unit: days] | 206 [1 to 18157] | 228 [23 to 3834] | 214 [1 to 18157]

OUTCOME MEASURES:

1. Primary Outcome: Complete Healing of the Study Ulcer by Week 16.
Time Frame: 16 weeks
Population: Intent-to-Treat population
Measure: Number; unit: participants
Arm/Group | Investigational Treatment (Dermagraft Plus Standard-of-Care) | Control (Standard-of-Care)
Number analyzed (Participants) | 274 | 263
participants | 201 | 176
Statistical Analysis 1: Comparison: Investigational Treatment (Dermagraft Plus Standard-of-Care) vs Control (Standard-of-Care); H0: the proportion of responders in the Dermagraft group = the proportion of responders in the Control group. HA: the proportion of responders in the Dermagraft group ≠ the proportion of responders in the Control group. The proportion of responders in the Dermagraft group was compared with the proportion of responders in the control group using the uncorrected chi-square test for 2x2 contingency tables. The difference between the groups was expected to be 13%; Test type: Superiority or Other; p = 0.1030, Chi-squared — This p-value did not meet the prespecified threshold for statistical significance of < 0.05; Unadjusted; Difference in proportions = 6.5

2. Secondary Outcome: Time-to-Complete Healing
Description: Kaplan-Meier survival analysis of the time to achieve median (50%) Complete Healing response in each treatment group.
Time Frame: From Week 0 visit to date subject's completely healed ulcer is 1st recorded as healed. If subject's ulcer not healed at 16 weeks, the "time until CH" was censored at 112 days.
Population: Intent-to-Treat population
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Investigational Treatment (Dermagraft Plus Standard-of=- Care): Weekly applications of Dermagraft and compression dressings, in combination with systematic surgical wound debridement.
Arm/Group | Investigational Treatment (Dermagraft Plus Standard-of=- Care) | Control (Standard-of-Care)
Number analyzed (Participants) | 274 | 263
days | 58 [36 to 113] | 64 [36 to 113]
Statistical Analysis 1: Comparison: Investigational Treatment (Dermagraft Plus Standard-of=- Care) vs Control (Standard-of-Care); Test type: Superiority or Other; p = 0.4046, Log Rank — This p-value did not meet the prespecified threshold for statistical significance of < 0.05; Median Difference (Final Values) = 6

3. Other Pre Specified Outcome: Complete Healing by Week 16: Ulcers <= 12 Months Duration
Time Frame: 16 weeks
Population: Pre-specified Subgroup of the Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | Investigational Treatment (Dermagraft Plus Standard-of-Care) | Control (Standard-of-Care)
Number analyzed (Participants) | 198 | 189
participants | 158 | 132
Statistical Analysis 1: Comparison: Investigational Treatment (Dermagraft Plus Standard-of-Care) vs Control (Standard-of-Care); Pre-specified subgroup analysis of the primary endpoint; Test type: Superiority or Other; p = 0.0239, Chi-squared — Unadjusted; Unadjusted; Difference in proportions = 10.0

ADVERSE EVENTS:
Arm/Group | Investigational Treatment (Dermagraft Plus Standard-of-Care) | Control (Standard-of-Care)
Serious Adverse Events (participants affected / at risk) | 28/274 | 24/263
Other Adverse Events (participants affected / at risk) | 168/274 | 157/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Treatment (Dermagraft Plus Standard-of-Care) (N=274) | Control (Standard-of-Care) (N=263)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrilation (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sick Sinus Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 3 (3) | 2 (2)
Drug intolerance (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 2 (2) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Facial bones fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Angiogram (Investigations) | 0 (0) | 1 (1)
Cardiac stress test (Investigations) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pupura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Implantable defibrilator replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Therapy regimen changed (Surgical and medical procedures) | 2 (2) | 0 (0)
Varicose vein operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Venous operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Treatment (Dermagraft Plus Standard-of-Care) (N=274) | Control (Standard-of-Care) (N=263)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 77 (77) | 60 (60)
Infected skin ulcer (Infections and infestations) | 22 (22) | 25 (25)
Excoriation (Injury, poisoning and procedural complications) | 20 (20) | 16 (16)
Hypertension (Vascular disorders) | 14 (14) | 13 (13)
Nasopharyngitis (Infections and infestations) | 18 (18) | 18 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (17) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Company-specific confidentiality agreement